CLINICAL TRIAL: NCT04304326
Title: Compare the Effectiveness of Functional Training Versus Resistance Exercises in Patients With Psoriatic Arthritis in Improving Functional Capacity, Disease Activity and Quality of Life
Brief Title: Comparison of the Effectiveness of Functional Training Versus Resistance Exercises in Patients With Psoriatic Arthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Principal Investigator, Diego Roger Silva, Principal investigator, Federal University of São Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 0928/2019
Record Dates: First submitted 2020-03-09; First posted 2020-03-11 (Actual); Last update posted 2023-03-29 (Actual); Status verified 2023-03

CONDITIONS: Psoriatic Arthritis
Keywords: Functional training; Physical exercise; Psoriatic arthritis; Quality of life
MeSH Terms: conditions — Arthritis, Psoriatic; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Single (Outcomes Assessor)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervational (Experimental): FT: Functional training with elastic band Underwent resistance exercise twice a week, for twelve weeks for the following muscles group: upper limbs, lower limbs and trunk.
  It was carried out two exercises for major muscle groups and one exercise for small muscles. The exercises were divided in 3 sets of 12 repetitions for each muscle group.
  The exercise program involved pectoral exercises: crucifix and seat supine; biceps: alternated screw; triceps: triceps pulley; back: standing handsaw and pulled ahead; quadriceps: leg extensor and finally gluteus: standing hips extension.
  Interventions: Other: Resistence Exercise
- Arms and Interventions (Experimental): Resistance exercise with weight training machines. Underwent resistance exercise twice a week, for twelve weeks for the following muscles group: upper limbs, lower limbs and trunk.
  It was carried out two exercises for major muscle groups and one exercise for small muscles. The exercises were divided in 3 sets of 12 repetitions for each muscle group. The intensity of the exercises was 60% of one-maximum repetition (1RM).
  The exercise program involved pectoral exercises: crucifix and seat supine; biceps: alternated screw; triceps: triceps pulley; back: standing handsaw and pulled ahead; quadriceps: leg extensor and finally gluteus: standing hips extension.
  Interventions: Other: Resistence Exercise

INTERVENTIONS:
Other: Resistence Exercise — Underwent resistance exercise twice a week, for twelve weeks for the following muscles group: upper limbs, lower limbs and trunk.
  It was carried out two exercises for major muscle groups and one exercise for small muscles. The exercises were divided in 3 sets of 12 repetitions for each muscle group. The intensity of the exercises was 60% of one-maximum repetition (1RM).
  The exercise program involved pectoral exercises: crucifix and seat supine; biceps: alternated screw; triceps: triceps pulley; back: standing handsaw and pulled ahead; quadriceps: leg extensor and finally gluteus: standing hips extension.

SUMMARY:
The aim of this study was to assess the effectiveness of Functional training versus resistance training in improving functional capacity, muscle strength, quality of life and disease activity in patients with PSA.

DETAILED DESCRIPTION:
The Functional Training Group (FT) used elastic bands and the Resistance Exercise Group (RE) used weight training machines. The FT patients performed functional training and RE performed resistance exercises for the following muscles group: upper limbs, lower limbs and trunk. It was used a machine "leg extension" for the training on the lower limbs. For upper limbs the investigators used a pulley triceps machine and front pull in addition to free weights (dumbbells).

In order to perform the exercise program, the study followed all the recommendations established by the American College of Sports Medicine (ACSM) (Ratamess et al., 2009). It was carried out two exercises for major muscle groups and one exercise for small muscles. The exercises were divided in 3 sets of 12 repetitions for each muscle group. The intensity of the exercises was 60% of one-maximum repetition (1RM).

The exercise program involved pectoral exercises: crucifix and seat supine; biceps: alternated screw; triceps: triceps pulley; back: standing handsaw and pulled ahead; quadriceps: leg extensor and finally gluteus: standing hips extension.

The patients were instructed to maintain their daily activities and to avoid any other nonpharmacological treatment.

ELIGIBILITY:
Inclusion Criteria:

Confirmed diagnosis of psoriatic arthritis, according to the CASPAR criteria

* Between 18 and 65 years of age, of both genders who agreed and signed the consent form.
* Patients should be-modifying drugs (DMARDs) on stable doses for at least three months and doses of non-steroidal anti-inflammatory drugs and corticosteroids stable for at least 4 weeks

Exclusion Criteria:

* Patients were excluded:

  * Uncontrolled cardiovascular disease
  * Decompensated diabetes mellitus; diseases
  * Severe psychiatric
  * Fibromyalgia
  * Other medical conditions that most disabling EA
  * History of regular exercise (at least 30 minutes 2 times per week) during the last 6 months
  * Arthroplasties of the hip and / or knee in the last 12 months; AND
  * Any other medical condition that prevents the patient from performing resistance exercises

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2020-07-30 (Actual)

PRIMARY OUTCOMES:
Change in the functional capacity | Baseline, after 45 and 90 days
  Evaluated by HAQ-S Health Assessment Questionnaire for the Spondyloarthropathies. There are 20 questions where the score ranges from zero to three. The higher the score, the greater the degree of functional impairment of the patient.

SECONDARY OUTCOMES:
Change in the quality of life | Baseline, after 45 and 90 days
  Evaluated by the SF-36 questionnaire; The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale, where the higher the score the less disability.

CONTACTS AND LOCATIONS:
Overall Officials: Jamil Natour, PHD, Study Chair — Federal University of São Paulo
Locations (1):
- São Paulo Hospital, São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Silva DR, Meireles SM, Brumini C, Natour J. Effectiveness of functional training versus resistance exercise in patients with psoriatic arthritis: randomized controlled trial. Adv Rheumatol. 2023 Dec 13;63(1):58. doi: 10.1186/s42358-023-00342-y. PMID 38093394